CLINICAL TRIAL: NCT02125695
Title: A Pilot Study to Evaluate Using Tape Harvesting to Collect Ribonucleic Acid From the Upper Epidermis of Healthy Volunteers and Subjects With Discoid Lupus, Subjects With Subacute Cutaneous Lupus, and Subjects With Atopic Dermatitis
Brief Title: Pilot Tape Harvesting Study
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 999LE003
Record Dates: First submitted 2014-04-25; First posted 2014-04-29 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Atopic Dermatitis; Healthy; Discoid Lupus Erythematosus; Subacute Cutaneous Lupus Erythematosus
MeSH Terms: conditions — Dermatitis, Atopic; Lupus Erythematosus, Discoid; Lupus Erythematosus, Cutaneous | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Specimens collected from skin taping and blood sampling.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy Volunteers: Skin taping; blood sampling; optional biopsy
  Interventions: Procedure: Skin Taping; Procedure: Blood Sampling; Procedure: Skin Biopsy
- Cutaneous lupus erythematosus: This group consists of participants affected with lupus (DLE, SCLE). Skin taping; blood sampling; optional skin biopsy (DLE participants); required skin biopsy (SCLE participants)
  Interventions: Procedure: Skin Taping; Procedure: Blood Sampling; Procedure: Skin Biopsy
- Atopic dermatitis: Skin taping; blood sampling; optional skin biopsy
  Interventions: Procedure: Skin Taping; Procedure: Blood Sampling; Procedure: Skin Biopsy

INTERVENTIONS:
Procedure: Skin Taping — Skin taping from affected and unaffected sites (4 tape harvestings/area plus photograph of taping site)
Procedure: Blood Sampling — Sampling for biomarker and basic research in CLE and AD
Procedure: Skin Biopsy — As described in the treatment arm

SUMMARY:
The main objectives of the study are: To determine if RNA recovery from tape harvesting allows for the identification of a disease gene signature (e.g., interferon [IFN] signature for lupus) or other biomarkers that may differentiate affected from normal or unaffected skin; To determine if the lupus gene signature is differentially expressed in the epidermis from active discoid lupus erythematosus (DLE) or subacute cutaneous lupus erythematosus (SCLE) lesions when compared with unaffected skin from the same participants and from the skin of healthy volunteers (HVs); To determine if the atopic dermatitis (AD) gene signature is differentially expressed in the epidermis from active AD lesions when compared with unaffected skin from the same participants and from the skin of HVs; and To correlate the levels of transcripts of targeted genes in the skin by tape harvesting with those obtained from the blood.

DETAILED DESCRIPTION:
No study drug is administered as part of this study. All participants except healthy volunteers will be treated according to standard clinical practice.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy volunteers must be in good overall health as determined by the Investigator, based on medical history, physical examination (per standard dermatology practice), and vital signs.
* Subjects with lupus must present with active DLE or SCLE skin disease (with or without systemic manifestations of SLE, as defined by ≥4 out of 11 classification criteria for SLE).
* Subjects with AD must have been diagnosed by the Eichenfield revised criteria of Hanifin and Rajka, disease duration for at least 2 years before Screening and disease activity defined as Investigator's Global Assessment (IGA) score ≥3 at screening

Key Exclusion Criteria:

* History of severe allergic or anaphylactic reactions or history of allergic reactions likely to be exacerbated by tape harvesting (e.g., allergy to adhesives).
* Other unspecified reasons that, in the opinion of the Investigator, make the subject unsuitable for enrollment.

Key Exclusion Criteria for Healthy Volunteers

* History of any clinically significant medical condition, as determined by the Investigator, that may impact study analyses

Key Exclusion Criteria for Subjects with Discoid or Subacute Cutaneous Lupus:

* Evidence of skin conditions other than DLE or SCLE at the Day 1 Visit that, in the opinion of the Investigator, would interfere with the study execution or analysis.
* History of malignancy in the last 5 years (nonmelanoma skin cancer that is considered cured by the Investigator will not be exclusionary).

Key Exclusion Criteria for Subjects With Atopic Dermatitis:

* History of any clinically significant medical condition, other than AD, as determined by the Investigator, that may impact study analyses, including, but not limited to: History of human immunodeficiency virus; History of hepatitis C virus or hepatitis B virus infection; Symptoms of bacterial or viral infection (including skin infection) within 14 days prior to the Day 1 Visit; History of malignancy in the last 5 years (nonmelanoma skin cancer that is considered cured by the Investigator will not be exclusionary).
* Evidence of skin conditions other than AD at the Day 1 Visit that, in the opinion of the Investigator, would interfere with the study execution or analysis.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are enrolled at selected investigational sites in a standard clinical practice setting
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2014-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
RNA expression of genes suspected to be associated with skin disease in affected versus unaffected skin in participants with skin disease | Day 1
  Participants with skin disease include participants affected with cutaneous lupus erythematosus ([CLE] i.e., DLE or SCLE), SCLE, AD
RNA expression of genes suspected to be associated with skin disease in healthy skin from HVs versus affected skin from participants with skin disease | Day 1
Comparison of RNA expression of genes suspected to be associated with skin disease in healthy skin from HVs versus unaffected skin from participants with skin disease | Day 1
Correlation between expression levels obtained from tape harvesting and those obtained from blood samples for each identified gene | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Boston, Massachusetts, United States